CLINICAL TRIAL: NCT03028766
Title: A Phase I Trial of WEE1 Inhibition with Chemotherapy and Radiotherapy As Adjuvant Treatment, and a Window of Opportunity Trial with Cisplatin in Patients with Head and Neck Cancer
Brief Title: WEE1 Inhibitor with Cisplatin and Radiotherapy: a Trial in Head and Neck Cancer
Acronym: WISTERIA
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: University of Birmingham (Other)
Collaborators: AstraZeneca (Industry); Cancer Research UK (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: RG_15-139; 2015-003583-37 (EudraCT Number); ISRCTN76291951 (Registry Identifier: ISRCTN Registry)
Record Dates: First submitted 2017-01-04; First posted 2017-01-23 (Estimated); Last update posted 2024-09-19 (Actual); Status verified 2024-09

CONDITIONS: Hypopharynx Squamous Cell Carcinoma; Oral Cavity Squamous Cell Carcinoma; Larynx Cancer
MeSH Terms: conditions — Squamous Cell Carcinoma of Head and Neck; Laryngeal Neoplasms | interventions — adavosertib; Cisplatin; Radiotherapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Group A - Pre-operative (Experimental): Patients will receive the cohort specified dose of AZD1775 by mouth, twice a day for 3 days, commencing on days 1 and 8. Cisplatin 40mg/m2 IV delivered over 1 hour on day 8. Patients in this group will commence surgery within 42 days of commencing pre-operative chemotherapy.
  Interventions: Drug: AZD1775; Drug: Cisplatin
- Group B - Post-operative: (Experimental): Patients will received the cohort specified dose of AZD1775 by mouth, twice a day for 3 days on days 2, 9, 23 and 30. Cisplatin 40mg/m2 IV delivered over 1 hour on days 2, 9, 16, 23 and 30. Intensity Modulated Radiotherapy will be delivered 5 days a week (once daily, Monday to Friday) for 6 weeks commencing within 3 months of surgery.
  Interventions: Drug: AZD1775; Drug: Cisplatin; Radiation: Radiotherapy

INTERVENTIONS:
Drug: AZD1775 — AZD1775 is a potent, selective small molecule inhibitor of WEE1
Drug: Cisplatin — Chemotherapy drug
Radiation: Radiotherapy — Intensity Modulated Radiotherapy
  Other Names: IMRT
  Arms: Group B - Post-operative:

SUMMARY:
This trial is to determine what dose of a drug called AZD1775 can safely be given in combination with cisplatin before surgery and with chemo-radiotherapy after surgery in patients with Head and Neck Cancer. The Investigators will also get some preliminary information regarding the effectiveness of this combined treatment.

DETAILED DESCRIPTION:
Patients with head and neck cancer with high-risk features are at increased risk of relapse after surgery. Surgery, often followed by cisplatin chemotherapy and radiotherapy is currently the standard treatment offered. Whilst chemo-radiotherapy improves cure rates, outcomes remain poor, and treatment has a significant impact on quality of life. Chemotherapy has yet to find a definitive role prior to surgery. There is therefore an urgent need to develop more effective treatments which improve cure rates for this patient population.

The purpose of this trial is to see whether incorporating a drug called AZD1775 into the management of head and neck cancer offers the possibility of addressing these clinical issues. AZD1775 is a drug that has been shown to increase the effect of cisplatin and of radiotherapy when tested in the laboratory. The blood samples and tumour biopsies taken during the trial will be important in learning as much as possible about the effects of AZD1775 on the body and to investigate how the tumour might develop resistance to the drug.

The WISTERIA trial is for patients aged between 18 and 70 years with cancer of the oral cavity, larynx and hypopharynx who are to undergo surgery. Patients recruited to Group A must have accessible tumours for re-biopsy, whilst patients recruited to Group B will be at high risk of relapse after surgery.

The primary objective of this trial is to see what dose of AZD1775 can safely be given in combination with cisplatin before surgery (Group A) and with chemo-radiotherapy after surgery (Group B). The Investigators will also get some preliminary information regarding the effectiveness of this combined treatment. To find the safe and effective dose of AZD1775, different doses will be tested for each Group.

ELIGIBILITY:
Inclusion Criteria:

* Histologically confirmed diagnosis of oral, laryngeal or hypopharyngeal squamous cell carcinoma
* Multi-Disciplinary Team (MDT) recommendation for surgical resection with curative intent
* Eastern Cooperative Oncology Group (ECOG) performance status 0/1
* Age ≥18 to ≤70 years
* Creatinine clearance, measured by Glomerular Filtration Rate (GFR), ≥ 60 ml/min at baseline calculated using local practice calculation. If this is ≤ 60 ml/min then an isotopic GFR may be carried out and must be > 60 ml/min
* Acceptable cardiac function. If significant cardiac history, then required for patient to have Left Ventricular Ejection Fraction (LVEF) ≥55% by echocardiogram (ECHO) or Multiple Gated Acquisition Scan (MUGA, if ECHO is equivocal)
* Normal liver and bone marrow function:

  * Haemoglobin (Hb) ≥10.0 g/dL or ≥100 g/L
  * Absolute neutrophil count (ANC) ≥1.5 x 109/L
  * Absolute platelet count ≥100 x 109/L
  * Aspartate transaminase (AST) or alanine aminotransferase (ALT) ≤2.5 upper limit of normal (ULN)
  * Total bilirubin ≤1.5 ULN (except for patients with known Gilbert's syndrome)
* Male and female participants must agree to take appropriate measures to prevent pregnancy. Contraceptive measures should be used for 2 weeks prior to trial entry, during the trial and for at least 6 months after last receiving treatment. Acceptable methods of contraception include total abstinence (if this is the patient's usual and preferred lifestyle choice), tubal ligation, combined oral, transdermal or intra-vaginal hormonal contraceptives, medroxyprogesterone injections (e.g. Depo-Provera), copper-banded intra-uterine devices; hormone impregnated intra-uterine systems and vasectomised partners. All methods of contraception (with the exception of total abstinence) should be used in combination with the use of a condom by their male sexual partner for intercourse.

Inclusion criteria Group A - in addition to general criteria

* Accessible tumours for re-biopsy under local anaesthetic or via ultrasound guided biopsy

Inclusion criteria Group B - in addition to general criteria

* High-risk histopathological features after surgical resection, i.e. nodal extra-capsular spread and/or tissue resection margin <1 mm as agreed at MDT
* Patients who have previously registered to Group A can be considered for inclusion in Group B

Exclusion Criteria:

* Any previous treatment for the same cancer, or previous head and neck malignancy, apart from laser excision of carcinoma in situ, with minimal residual functional deficit or registration and treatment in Group A prior to surgery
* Patients with cancer of the oropharynx or non-primary cancer will not be included
* Any metastatic disease from any primary site
* Use of an Investigational Medicinal Product (IMP) concurrently or within 4 weeks of starting this trial
* Uncontrolled intercurrent illness, which will interfere with the patient's participation in the trial, e.g.:

  * myocardial infarction within 6 months
  * congestive cardiac failure
  * unstable angina
  * symptomatic cardiomyopathy
  * chronic infections
  * active peptic ulcer or liver disease
  * serious psychiatric condition limiting ability to comply with trial protocol
* Clinical evidence of current heart failure (≥New York Heart Association (NYHA) Class II)
* Clinical evidence of atrial fibrillation (with heart rate >100 bpm, within 6 months prior to trial entry)
* Unstable ischaemic heart disease (Myocardial Infarction within 6 months prior to trial entry or angina requiring the use of nitrates greater than once weekly)
* Patients who have a history of Torsades de pointes (unless all risk factors that contributed to Torsades de pointes have been corrected)
* Active gastro-intestinal disease that might limit absorption of study drug, e.g. coeliac disease, Crohn's disease, ulcerative colitis, pancreatic insufficiency
* Evidence of any psychological, familial, sociological or geographical condition potentially hampering protocol compliance
* Participation in another interventional clinical trial whilst taking part in this trial
* Patients who are unable to discontinue any prohibited drug and unable to tolerate a washout period for at least 14 days prior to trial entry
* Clinical judgement by the Investigator that the patient should not participate in the study
* Known hypersensitivity to the study drugs or active substances or excipients of the preparations
* Pregnant or breast feeding patients
* Significant pre-existing neuropathy which currently interferes with the patient's daily life
* Mean resting corrected QTc interval using the Fridericia formula (QTcF) >450 msec (male) and >470 msec (female) (as calculated per institutional standards) obtained from 3 electrocardiograms (ECGs) 2-5 minutes apart at study entry, or congenital long QT syndrome
* Inability to swallow oral medications

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 9 (Actual)
Dates: Start 2017-06-22 (Actual); Primary Completion 2019-10-31 (Actual); Study Completion 2021-02-03 (Actual)

PRIMARY OUTCOMES:
Recommended dose(s) of AZD1775 | Group A - Up to 42 days from start of treatment; Group B - Up to 12 weeks from the start of treatment
  Group A: The highest safe dose of AZD1775 in combination with cisplatin with a predefined target Dose Limiting Toxicity probability of 25% for up to 42 days from start of treatment.
  Group B: The maximum tolerated dose of AZD1775 in combination with cisplatin/radiotherapy with a target DLT of 30% for up to 12 weeks from the start of treatment.
Safety profile of AZD1775 for Group A and Group B by reporting of all Adverse Events, Serious Adverse Events, Suspected Unexpected Adverse Reactions, deaths, deviations and withdrawal as assessed by the Safety Committee. | From registration, while on treatment and during follow up periods
  Safety profile of AZD1775 in combination with cisplatin in Group A and cisplatin/radiotherapy in Group B.

SECONDARY OUTCOMES:
Disease-free survival in Groups A and B | Patients will be followed-up clinically for 12 weeks in Group A and for 12 months in Group B.
  Disease-free survival is defined as the time from trial entry to date of disease recurrence, progression or patient death until end of follow up period.

CONTACTS AND LOCATIONS:
Overall Officials: Hisham Mehanna, Principal Investigator — University of Birmingham
Locations (6):
- United Kingdom (6):
  - University Hospital Birmingham Nhs Foundation Trust, Birmingham, West Midlands
  - Beatson West of Scotland Cancer Centre, Glasgow
  - St. James' University Hospital, Leeds Teaching Hospital NHS Trust, Leeds
  - The Royal Marsden Hospital, London
  - University College London Hospitals, London
  - Clatterbridge Cancer Centre, Metropolitan Borough of Wirral

IPD SHARING:
Plan to Share IPD: Yes
The datasets generated during and/or analysed during the current study are available from the corresponding author on reasonable request. The CRCTU is committed to responsible and controlled sharing of anonymised clinical trial data with the wider research community to maximise potential patient benefit while protecting the privacy and confidentiality of trial participants. Data anonymised in compliance with the Information Commissioners Office requirements, using a procedure based on guidelines from the MRC Methodology Hubs, will be available for sharing with researchers outside of the trials team within 6 months of the primary publication. More detailed information on the CRCTU's Data Sharing Policy and the mechanism for obtaining data can be found on the CRCTU website: https://www.birmingham.ac.uk/research/activity/mds/trials/crctu/index.aspx.
Supporting Information: Study Protocol, SAP, ICF, Analytic Code
Time Frame: Data will be available within 6 months of the primary publication.
Access Criteria: See Plan Description above.

REFERENCES:
- [Background] Kong A, Kirkham AJ, Savage JS, Mant R, Lax S, Good J, Forster MD, Sacco JJ, Schipani S, Harrington KJ, Yap C, Mehanna H. Results and lessons learnt from the WISTERIA phase I trial combining AZD1775 with cisplatin pre- or post-operatively in head and neck cancer. BJC Rep. 2024;2(1):6. doi: 10.1038/s44276-023-00026-6. Epub 2024 Jan 29. PMID 39220748
- [Background] Kong A, Good J, Kirkham A, Savage J, Mant R, Llewellyn L, Parish J, Spruce R, Forster M, Schipani S, Harrington K, Sacco J, Murray P, Middleton G, Yap C, Mehanna H. Phase I trial of WEE1 inhibition with chemotherapy and radiotherapy as adjuvant treatment, and a window of opportunity trial with cisplatin in patients with head and neck cancer: the WISTERIA trial protocol. BMJ Open. 2020 Mar 16;10(3):e033009. doi: 10.1136/bmjopen-2019-033009. PMID 32184305
- See also: Trial Website — https://www.birmingham.ac.uk/research/crctu/trials/wisteria/index.aspx
- See also: ISRCTN (including basic results) — https://www.isrctn.com/ISRCTN76291951